CLINICAL TRIAL: NCT05007509
Title: A Phase I/IIa Study to Evaluate Safety and Immunogenicity of Recombinant Protein RBD Candidate Vaccine Against SARS-CoV-2 in Adult Healthy Volunteers
Brief Title: Safety and Immunogenicity Study of Recombinant Protein RBD Candidate Vaccine Against SARS-CoV-2 in Adult Healthy Volunteers (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laboratorios Hipra, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIPRA-HH-1; 2021-001411-82 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-08-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Covid19; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19 | interventions — KPNA1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 vaccine HIPRA (Experimental): Subjects will receive 2 injections of COVID-19 vaccine HIPRA administered 21 days apart.
  Interventions: Biological: COVID-19 vaccine HIPRA 10; Biological: COVID-19 vaccine HIPRA 20; Biological: COVID-19 vaccine HIPRA 40
- Commercial COVID-19 vaccine (Active Comparator): Subjects will receive 2 injections of commercial COVID-19 vaccine administered 21 days apart.
  Interventions: Biological: Commercial COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine HIPRA 10 — One sentinel subject and 4 additional subjects will be assigned to COVID-19 vaccine HIPRA 10 µg
  Other Names: COHORT 1
  Arms: COVID-19 vaccine HIPRA
Biological: COVID-19 vaccine HIPRA 20 — One sentinel subject and 9 additional subjects will be assigned to COVID-19 vaccine HIPRA 20 µg
  Other Names: COHORT 2
  Arms: COVID-19 vaccine HIPRA
Biological: COVID-19 vaccine HIPRA 40 — One sentinel subject and 9 additional subjects will be assigned to COVID-19 vaccine HIPRA 40 µg
  Other Names: COHORT 3
  Arms: COVID-19 vaccine HIPRA
Biological: Commercial COVID-19 vaccine — One subject in cohort 1 and 2 subjects in Cohort 2 and 3 will be assigned to Commercial COVID-19 vaccine
  Arms: Commercial COVID-19 vaccine

SUMMARY:
This is a first-in-human, phase I/IIa, randomized, controlled, observer-blinded, dose-escalation, multicentre clinical trial to evaluate safety and immunogenicity of COVID-19 HIPRA vaccine in adult healthy volunteers.

DETAILED DESCRIPTION:
The study population includes 30 healthy adults aged 18-39 which will be distributed in 3 cohorts, receiving three different doses of antigen, 10 µg, 20 µg and 40 µg. In each cohort, patients will be randomized in ratio of 10:2 test:commercial vaccine, following an staggered enrolment with a sentinel subject in each cohort. Each participant will receive 2 immunisations separated by 21 days, and will be followed for 48 weeks after the second dose

ELIGIBILITY:
Inclusion Criteria:

* Adults males or females between 18-39 years of age at the day of screening.
* Willing and able to comply with scheduled visits, laboratory test, complete diaries and other study procedures.
* Body Mass Index 18 to 40 Kg/m2 at screening.
* COVID19 negative PCR test and negative serum IgG binding antibody response to the SARS-CoV-2 S glycoprotein at screening or prior the first vaccination.
* Willing to avoid all other vaccines within 4 weeks before and after each injection. Seasonal influenza vaccination is allowed if it is received at least 14 days before or after the vaccination.
* Women of childbearing potential must have a negative pregnancy test in urine before the inclusion of the study and prior to each vaccination.
* If female of childbearing potential, willing to use highly effective contraceptive methods or have practiced sexual abstinence from the screening visit until 8 weeks after the last injection.
* If male and not sterilized, willing to avoid impregnating female partners from screening until 18 weeks after last injection.
* Willing and able to provide written informed consent prior the initiation of any study procedures.

Exclusion Criteria:

* Pregnant or lactating or intending to become pregnant or plans to breastfeed during the study.
* Positive pregnancy test at screening or prior to each vaccination.
* Any medical disease (acute, subacute, intermittent or chronic) or condition that in the opinion of the investigator compromise the volunteer's safety, preclude vaccination or compromise interpretation of the results.
* History of serious psychiatric condition likely to affect participation in the study (e-g- ongoing severe depression, history of admission to an in-patient psychiatric facility, recent suicidal ideation, history of suicide attempt, bipolar disorder, personality disorder, alcohol and drug dependency, severe eating disorder, psychosis, use of mood stabilisers or antipsychotic medication).
* History of respiratory disease (e.g., chronic obstructive pulmonary disease (COPD) and asthma) requiring any daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years.
* History of significant cardiovascular disease including hypertension (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
* History of neurological or neurodevelopmental conditions (e.g., migraines, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).
* Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections.
* Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital).
* Acute illness within 72 hours prior each vaccination that in the opinion of the investigator may interfere the evaluation of safety parameters.
* Usage of any investigational drug ≤ 90 days prior to study entry or plan to participate in another research involving an investigational product (drug/biologic/device) within 12 months after the first study vaccination.
* History of hypersensitivity or severe allergic reaction including anaphylaxis, generalized urticarial, angioedema and other significant reactions related to food, drugs, vaccines or pharmaceutical agents.
* History of allergic disease or reactions likely to be exacerbated by any component of the COVID-19 vaccine HIPRA.
* Use of any immunosuppressant, glucocorticoids, or other immune-modifying drugs within 2 months prior to first study vaccination; or anticipation of the need for immunosuppressive treatment within 6 months after last vaccination.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days prior to first study vaccination.
* Known disturbance of coagulation (iatrogenic or congenital) or blood dyscrasias.
* Known bleeding disorder (e-g- factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
* Chronic liver disease.
* Positive test for HIV types 1 or 2 infection, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV Abs) at screening.
* Suspected or known current alcohol abuse or any other substances abuse (except tobacco).
* History of COVID-19 infection.
* Receipt of medications intended to prevent COVID-19.
* Ever received an experimental vaccine against COVID-19.
* Close contact of anyone known to have SARS-CoV-2 infection within 15 days prior to screening visit.
* Being directly involved in the conduct of the study.
* Any condition and/or laboratory finding that at the investigator consideration would interfere with the study or put at risk the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number and percentage of solicited local and systemic reactogenicity adverse events for 7 days following each vaccination. | 7 days
Number and percentage of unsolicited local and systemic reactogenicity adverse events for 28 days following each vaccination. | 28 days

SECONDARY OUTCOMES:
Change from baseline in hematology and biochemistry laboratory values at 7 days following each vaccination | 7 days
Number and percentage of serious adverse events throughout the study duration. | 357 days
Number and percentage of adverse events of special interest (AESI) throughout the study | 357 days
Number and percentage of medically attended adverse events (MAAE) related to study vaccine throughout the study duration | 357 days
Neutralization titer measured as Inhibitory concentration 50 (IC50) for each individual sample and geometric mean titer (GMT) for group comparison at Day 21 and 35 | Day 21 and 35
Geometric mean fold rise (GMFR) in neutralizing antibodies titers from baseline at Day 21 and 35. | Day 21 and 35
Neutralization titer measured as IC50 for each individual sample and GMT for group comparison at 24 and 48 weeks after the second dose | week 27 and week 51
GMFR in neutralizing antibodies titers from baseline at 24 and 48 weeks after the second dose. | week 27 and week 51
Binding antibody IgG titer measured for each individual sample and GMT for group comparison at Day 21 and 35 | Day 21 and 35
GMFR in IgG titer from baseline at Day 21 and 35 | Day 21 and 35
Binding antibody IgG titer measured for each individual sample and GMT for group comparison at 24 and 48 weeks after the second dose. | week 27 and week 51
GMFR in IgG titer from baseline at 24 and 48 weeks after the second dose | week 27 and week 51
T-cell-mediated response to the SARS-CoV-2 S protein as measured by whole PBMC stimulation by ELISpot at baseline and at Day 35. | Day 35
CD4+/CD8+ T-cell response to the SARS-CoV-2 S protein as measured by in vitro PBMC stimulation by cytokine staining assays at baseline and at Day 35 | Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Elia Torroella, Study Chair — Laboratorios Hipra, S.A.
Locations (2):
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Dr. Josep Trueta, Girona

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Derived] Leal L, Pich J, Ferrer L, Nava J, Marti-Lluch R, Esteban I, Pradenas E, Raich-Regue D, Prenafeta A, Escobar K, Pastor C, Ribas-Aulinas M, Trinite B, Munoz-Basagoiti J, Domenech G, Clotet B, Corominas J, Corpes-Comes A, Garriga C, Barreiro A, Izquierdo-Useros N, Arnaiz JA, Soriano A, Rios J, Nadal M, Plana M, Blanco J, Prat T, Torroella E, Ramos R; HIPRA-HH-1 study group. Safety and immunogenicity of a recombinant protein RBD fusion heterodimer vaccine against SARS-CoV-2. NPJ Vaccines. 2023 Sep 29;8(1):147. doi: 10.1038/s41541-023-00736-5. PMID 37775521